CLINICAL TRIAL: NCT07405034
Title: Artificial Intelligence Driven Exercises Versus Conventional Exercises Therapy for Patellofemoral
Brief Title: AI Driven EX Versus Conventional in PFPS
Acronym: AI- PFPS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa hamdi elsaid rizk, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/006096
Record Dates: First submitted 2026-01-26; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Patello Femoral Pain Syndrome

STUDY DESIGN:
Intervention Model Description: This study is randomized controlled trial and includes 40 participants .These participants divided into 2 groups (A, B), each group will be assessed with 3 measurments (vas ,dynamic knee valgus, Kujala Anterior Knee Pain Scale) and each group will receive difeerent treatments.
  The individuals in group A(study group) will preceive AI driven exercises program while the individual in group B will receive conventional exercises therapy program. Participants in the both groups are prescribed a 6-week comprehensive exercises program (3 sessions per week) day after day and assessment procedure will be performed pre and post treatmeant .
Who Masked: Participant
Masking Description: All participants will randomized via random generator (www.randomization.com). All patients will be blinded to group allocation by ensuring that they will be unaware of the exercises performed by the other group. To maintain the blinding, the intervention sessions will be delivered separately to members of each treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ( AI driven EX for study group ) (Active Comparator): The individuals in group A(study group) will preceive AI driven exercises program while the individual in group B will receive conventional exercises therapy program. Participants in the both groups are prescribed a 6-week comprehensive exercises program (3 sessions per week) day after day and assessment procedure will be performed pre and post treatmeant
  Interventions: Other: Ai driven EX
- conventional ex group (Other): The individual in group B will receive conventional exercises therapy program. Participants in the both groups are prescribed a 6-week comprehensive exercises program (3 sessions per week) day after day and assessment procedure will be performed pre and post treatmeant .
  Interventions: Other: conventional exercises therapy program

INTERVENTIONS:
Other: conventional exercises therapy program — The individual in group B will receive conventional exercises therapy program. Participants are prescribed a 6-week comprehensive exercises program (3 sessions per week) day after day and assessment procedure will be performed pre and post treatmeant
  Arms: conventional ex group
Other: Ai driven EX — The individuals in group A(study group) will preceive AI driven exercises program . Participants in the both groups are prescribed a 6-week comprehensive exercises program (3 sessions per week) day after day and assessment procedure will be performed pre and post treatmeant
  Arms: ( AI driven EX for study group )

SUMMARY:
This study aims to investigate and compare the effect of AI driven exercises program versus the conventional exercises therapy program on pain, function and dynamic knee valgus angle in treatment of patellofemoral pain syndrome.This study is randomized controlled trial and includes 40 participants .These participants divided into 2 groups (A, B), each group will be assessed with 3 measurments (vas ,dynamic knee valgus, Kujala Anterior Knee Pain Scale) and each group will receive difeerent treatments.

The individuals in group A(study group) will preceive AI driven exercises program while the individual in group B will receive conventional exercises therapy program. Participants in the both groups are prescribed a 6-week comprehensive exercises program (3 sessions per week) day after day and assessment procedure will be performed pre and post treatmeant .

DETAILED DESCRIPTION:
PURPOSE : This study aims to investigate and compare the effect of AI driven exercises program versus the conventional exercises therapy program on pain, function and dynamic knee valgus angle in treatment of patellofemoral pain syndrome.

BACKGROUND:

Patellofemoral pain syndrome (PFPS) is one of the most common knee problems that disturb function and daily activities (Menek et al .,2025). Symptoms of PFPS can develop either slowly or abruptly, and pain tends to worsen with activities such as squatting, prolonged sitting, stair climbing, jumping, or running (Menek et al .,2025). PFPS affects approximately 25% of physically active individuals (Smith et al .,2018).

Core training significantly improves pain and functional limitations in patients with PFP and improves lower extremity motor performance to some extent (Y. Wang et al., 2024). These results draw more attention to the importance of the core muscle performance for both prevention and rehabilitation of the knee injuries

HYPOTHESES:

A-Primary Hypotheses:

This study will hypothesize that:

1. There will be no significant effect of AI driven exercises program on pain in treatment of patients PFPS .
2. There will be no significant effect of AI driven exercises program on function in treatment of patients PFPS .
3. There will be no significant differences of AI driven exercises program and on dynamic knee valgus in treatment of patients PFPS.
4. There will be no significant differences of conventional exercises therapy on pain in treatment of patients PFPS.
5. There will be no significant differences of conventional exercises therapy on function in treatment of patients PFPS.
6. There will be no significant differences of conventional exercises therapy dynamic knee valgus in treatment of patients PFPS.

RESEARCH QUESTION:

This study will try to answer the following questions:

This study will try to answer:What are the effects of of AI driven exercises program and the conventional exercises therapy program on pain, function and dynamic knee valgus angle in treatment of patellofemoral pain syndrome ?

ELIGIBILITY:
Inclusion Criteria:

* Their ages range from 18- 40 years old, including both genders (male & female).
* Their BMI will be ≤ 29 kg/m2.
* A traumatic knee pain persisting for at least three months.

Exclusion Criteria:

* Any congenital deformity of the lower limb,
* Any recent injuries and surgeries
* severe foot deformities such as hallux valgus and claw toe
* Neuromuscular and neurological disorders.- history of patellofemoral dislocation, subluxation .

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02-26 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Kujala Anterior Knee Pain Scale | up to 6 weeks
  a 13-item scale assessing knee functionality. The total Kujala score ranges from 0 to 100, with higher values indicating better performance. Additionally, The Kujala score is known for its reliability and validity in assessing patients with frozen PFPS

SECONDARY OUTCOMES:
visual analog scale | up to 6 weeks
  Pain intensity is assessed using the visual analog scale. Participants are instructed to indicate their pain level on a line ranging from 0 to 10, with 0 representing no pain and 10 indicating unbearable pain

CONTACTS AND LOCATIONS:
Overall Officials: SALWA FADL abdelmegeed, Professor of Physical Therapy, Study Director — Cairo University
Locations (2):
- Egypt (2):
  - the out-patient clinic faculty of physical therapy, Cairo University,, Cairo, The Capital
  - the out-patient clinic faculty of physical therapy, Cairo University,, Cairo

IPD SHARING:
Plan to Share IPD: No
Data is available with correspondig offer on reasonable request